CLINICAL TRIAL: NCT04699643
Title: A Phase I/II Study of FGFR4 Inhibitor EVER4010001 in Combination With PD-1 Inhibitor Pembrolizumab in Patients With Advanced Solid Tumors With Dose Escalation and Expansion to Selected Indications
Brief Title: FGFR4 Inhibitor EVER4010001 in Combination With PD-1 Inhibitor Pembrolizumab in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EverNov Medicines (Zhuhai Hengqin) Co., Ltd (Industry)
Collaborators: Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVER401-001
Record Dates: First submitted 2020-12-29; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EVER4010001 combination with Pembrolizumab (Experimental): EVER4010001 combination with Pembrolizumab, EVER4010001 started dose escalation from 40mg bid, and then to 60mg bid, 80mg bid, 100mg bid and 120 mg bid if applicable, dose escalation decision will be made by safety monitoring committee which is composed of the study team members. After phase II dose was recommended by safety monitoring committee, this dose will be applied to phase II patients. Pembrolizumab will be administered at 200mg every 3 weeks through the study.
  Interventions: Drug: EVER4010001

INTERVENTIONS:
Drug: EVER4010001 — Please refer to information in arm/group descriptions.
  Other Names: Pembrolizumab

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of EVER4010001 in combination with Pembrolizumab in Patients with Advanced Solid Tumors. And in phase II to assess the anti-tumor efficacy of EVER4010001 in combination with Pembrolizumab in treating selected indications using appropriate biomarkers.

DETAILED DESCRIPTION:
This is a phase I/II, single arm, multicenter study of EVER4010001 combination with Pembrolizumab in advanced solid tumor patients. The primary endpoint of phase I will be Dose-limiting toxicities (DLTs) observed in combined administration of EVER4010001 and Pembrolizumab. And the primary endpoint of phase II will be the ORR per RECIST v1.1 in all treated patients.

Patients will be treated until progression requiring discontinuation of further treatment, unacceptable toxicity, study withdrawal, or death, whichever comes first. Tumor response and progression will be assessed using RECIST v1.1 and assessment by investigator at the trail center will be sufficient for decisions on continuation of treatment. All patients will visit the investigator at regular intervals for assessment of safety parameters and AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any procedures that are related to this study.
2. Patients (male or female) ≥ 18 years of age
3. Eastern Cooperative Oncology Group (ECOG) performance status≤1
4. Presence of at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
5. Phase I study part: Histologically or cytologically confirmed metastatic or locally advanced solid tumors, for which no standard therapy exits or the standard therapy has failed.

Phase II study part: 1. Histologically or cytologically confirmed metastatic or locally advanced solid tumors of the selected indications. 2. Positive FGF19 in IHC test results of tumor tissues in pre-screening.

Exclusion criteria:

1. Prior therapies within the following time frames prior to the first dose of study treatment:

   * Last dose of conventional cytotoxic chemotherapy: ≤4 weeks ((≤ 6 weeks for nitrosoureas and mitomycin-C);
   * Drugs with anti-tumor activity (e.g., antibodies): ≤4 weeks
   * Non-cytotoxic small molecule therapeutics (e.g., sorafenib): ≤5 half-lives or ≤2 weeks (whichever is longer)
   * Previous wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 4 weeks and limited field radiation for palliation ≤ 2 weeks (including particle implantation such as I125);
   * Participation in a prior investigational study: ≤ 4 weeks;
   * Drugs with immunomodulatory activity (such as thymosin, interferon, interleukin, etc.) ≤ 6 weeks.
2. Major surgery within 4 weeks of receiving the first dose of study treatment (mediastinoscopy, insertion of a central venous access device and insertion of a feeding tube are not considered major surgery).
3. Subject having out of range laboratory values including hematology, chemistry and coagulation indicators. See Section 5.3 for specific indicators.
4. Use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GM-CSF, M CSF), blood transfusion products (e.g., whole blood, plasma, apheresis platelets, etc.), thrombopoietin mimetics or erythroid stimulating agents ≤ 2 weeks prior to start of study treatment. If erythroid stimulating agents were initiated more than 2 weeks prior to the first dose of study treatment and the patient is on a stable dose, they can be maintained.
5. Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 5 years prior to study entry; completely resected basal cell and squamous cell skin cancers and completely resected carcinoma in situ of any type.
6. Symptomatic CNS metastases which are neurologically unstable, or CNS metastases requiring local CNS directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids within 2 weeks of first dose of study treatment.
7. Serous effusion with clinically significant symptoms (such as shortness of breath, abdominal distention, etc.).
8. Major acute or chronic infections, including:

   1. Positive human immunodeficiency virus (HIV) antibody screening or known acquired immunodeficiency syndrome (AIDS);
   2. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection: positive HBV-DNA copies (>2000 IU/mL) and/or other activity indicators; positive HCV antibody and HCV-RNA test result;
   3. active TB (such as exposure history or positive TB test; AND clinical symptoms, physical or imaging manifestations);
   4. Ongoing antibiotic treatment of serious acute infections.
9. Previous treatment with a selective FGF19-FGFR4 targeted therapy and/or pan-FGFR inhibitor.
10. Patients receiving treatment with cytochrome P450 (CYP)1A2, CYP2C9 and CYP3A4/5 substrates with a narrow therapeutic index (NTI) that cannot be discontinued for the duration of the study.
11. Patients receiving known BSEP efflux transporter inhibitors that cannot be discontinued 3 days prior to the start of study treatment and during the course of the study.
12. Current evidence of calcium-phosphate homeostasis impairment. See Section 5.3 for specific indicators.
13. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral EVER4010001 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, small bowel resection).
14. Ongoing active diarrhea requiring medications (e.g. bile acid sequestrant (BAS), loperamide).
15. Irritable bowel syndrome with signs/symptoms or requires medications.
16. Any previous specific target T cell co-stimulation or immune checkpoint pathway treatment, including but not limited to PD-1 inhibitors, PD-L1 / 2 inhibitors or other targeted T cell drugs.
17. Use of systemic chronic steroid therapy (≥ 10mg/day prednisone or equivalent) or any immunosuppressive therapy two weeks prior to start of study treatment. Topical, inhaled, nasal and ophthalmic steroids are allowed.
18. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment (except inactivated seasonal influenza vaccines).
19. Active known or suspected autoimmune disease. Patients with vitiligo, residual hypothyroidism only requiring hormone replacement, or psoriasis not requiring systemic treatment can be included.
20. History of severe hypersensitivity reactions to any ingredient of study treatment and other monoclonal antibodies (mAbs) and/or their excipients.
21. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

    -Clinically significant or uncontrolled heart disease such as congestive heart failure requiring treatment (New York Heart Association Grade ≥ 2), uncontrolled hypertension (defined by Systolic Blood Pressure > 160 mmHg/ Diastolic Blood Pressure > 100mmHg (average of three consecutive readings) at rest despite medical treatment, clinically significant arrhythmia; QTcF > 470 msec on screening ECG or congenital long QT syndrome; acute myocardial infarction or unstable angina pectoris < 3 months prior to screening.
22. History of liver or other organ transplantation.
23. History of interstitial lung disease or pneumonia requiring oral or intravenous steroids.
24. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
25. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing with study treatment and for the following duration after discontinuation of study treatment: See Section 5.3 for specific contraception methods.
26. Sexually active males unless they use a condom during intercourse while receiving study treatment and for the following period after the last dose of study treatment, and should not father a child in this period.
27. Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures. Any severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) observed in combined administration of EVER4010001 and Pembrolizumab | up to 12 months
  Dose-limiting toxicities (DLTs) observed in combined administration of EVER4010001 and Pembrolizumab
Objective response rate (ORR) by IRC according to RECIST v 1.1 | 3 years
  Objective response rate (ORR) by IRC according to RECIST v 1.1

SECONDARY OUTCOMES:
PK parameters of EVER4010001: maximum observed concentration (Cmax) | 3 years
  PK parameters of EVER4010001: maximum observed concentration (Cmax)
Objective response rate (ORR) | 3 years
  Objective response rate (ORR)
Disease control rate (DCR) | 3 years
  Disease control rate (DCR)
Duration of response (DOR) | 3 years
  Duration of response (DOR)
Adverse events (AEs) and serious adverse events (SAEs) defined by National Cancer Institute-Common terminology criteria for adverse events (NCI-CTCAE) v5.0 | 3 years
  Adverse events (AEs) and serious adverse events (SAEs) defined by National Cancer Institute-Common terminology criteria for adverse events (NCI-CTCAE) v5.0
Exploratory biomarkers include Total bile acids, 7-α-hydroxy-4-cholesten-3-one (C4), circulating FGF19, etc. | 3 years
  Exploratory biomarkers include Total bile acids, 7-α-hydroxy-4-cholesten-3-one (C4), circulating FGF19, etc.
Progression-free survival (PFS) | 3 years
  Progression-free survival (PFS)
Overall survival (OS) | 3 years
  Overall survival (OS)
Immunogenicity of Pembrolizumab: anti-drug antibody (ADA) | 3 years
  Immunogenicity of Pembrolizumab: anti-drug antibody (ADA)
FGF19 expression in tumor cells and tumor microenvironment cells by immunohistochemical testing | 3 years
  FGF19 expression in tumor cells and tumor microenvironment cells by immunohistochemical testing
PK parameters of EVER4010001: area under the concentration-time curve (AUC) | 3 years
  PK parameters of EVER4010001: area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Principal Investigator — Department of Gastrointestinal Oncology, the Fifth Medical Center, Chinese PLA General Hospital
Locations (1):
- Department of Gastrointestinal Oncology, the Fifth Medical Center, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No